CLINICAL TRIAL: NCT03719599
Title: Cross-Sectional Survey of Plasmodium and Other Parasites in Pregnant Women and Children Around Margibi and Montserrado Counties, Liberia
Brief Title: Plasmodium and Other Parasites in Pregnant Women and Children Around Margibi and Montserrado Counties, Liberia
Status: Completed | Type: Observational
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 999919007; 19-I-N007
Record Dates: First submitted 2018-10-24; First posted 2018-10-25 (Actual); Last update posted 2025-11-20 (Actual); Status verified 2025-04-03

CONDITIONS: Malaria
Keywords: Malaria; Infection; Seasonal; Parasitemia; Organism; Natural History
MeSH Terms: conditions — Malaria; Infections; Parasitemia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Children: Children 6 -12 months of age presenting for routine clinic visits
- Pregnant Women: Pregnant Women 18 years and older presenting for routine clinic visits

SUMMARY:
Background:

The disease malaria affects many people in Liberia and other parts of Africa. It is caused by germs that are spread by mosquito bites. It may be mild but can be serious or can lead to death if not diagnosed and treated. Children younger than 5 years old and pregnant women are most at risk of malaria. Worms also infect many people in Liberia. They can be caused by mosquito bites or by touching soil or still water. Worm infections can be mild or serious. Doctors in Liberia and their NIH partners want to learn more about these diseases in women and children.

Objective:

To measure how much malaria and worm infections there are in pregnant women and children in two counties of Liberia.

Eligibility:

Pregnant women ages 18 and older and children ages 6 12 months seeking routine care at C.H. Rennie Hospital or the Duport Road Health Center

Design:

Participants will be screened with questions about their health or their child s health.

Participants will be asked further questions about their health and about their home life.

Participants will give a small amount of blood by finger prick. This will be tested to see if they have malaria or some types of worms, and for research studies.

Participants who are sick from malaria will be treated at a study clinic. Treatment will follow standards of the Liberia and/or the World Health Organization.

DETAILED DESCRIPTION:
Malaria caused by Plasmodium falciparum continues to be a global problem with devastating consequences, in particular for at-risk populations such as pregnant women and young infants. Pregnancy malaria is associated with low birth weight (LBW), maternal anemia, and gestational hypertension; both inflammation and the fetal response to infection may contribute to these poor outcomes. Placental malaria (PM) is caused by P. falciparum-infected erythrocytes that bind to the placental receptor chondroitin sulfate A (CSA) and sequester in the placenta, where they cause disease and may lead to death of the mother and her offspring. Women become resistant to PM as they acquire antibodies that target surface proteins of placental parasites. In areas of stable transmission, acute severe malaria syndromes are limited to children under 5 years of age. The pathogenesis of severe malaria remains poorly understood, although some evidence suggests that parasites causing severe malaria may express distinct antigens on the surface of infected erythrocytes. Thus, vaccines to prevent malarial disease may need to target distinct antigens in order to protect pregnant women or young children.

The primary hypothesis in this study is that the burden of P. falciparum infection around Margibi and Montserrado is sufficient to support future studies of malaria pathogenesis and immunity. In addition to assessing malaria burden this study will build up diagnostic laboratory capacity for malaria diagnostics. We plan to enroll 2920 pregnant women and 2920 children (6-12 months of age) into a cross sectional study that will be conducted in Margibi and Montserrado counties, Liberia. Women presenting for routine antenatal visits and presenting for well-baby clinic visits (e.g. vaccinations, vitamins) at C.H. Rennie Hospital in Margibi or Duport Road Health Center in Montserrado will be enrolled. Samples collected from the women and children will be examined for evidence of infection by Plasmodium and other parasitic diseases in order to assess prevalence in this key reservoir population. For our primary outcome, we will determine the prevalence of P. falciparum infection in these two key demographic groups, including their annual and seasonal variations, as these data will form the basis to design future natural history or interventional studies at these sites. For our secondary outcomes, we will determine the prevalence of other parasitic diseases, such as filaria, S. stercoralis, and schistosomes by serologic assays of blood samples.

ELIGIBILITY:
* INCLUSION CRITERIA:
* For pregnant women, a study participant must satisfy the following criteria to be enrolled in this study:

  * Pregnant woman >=18 years of age reporting for routine care at the center without acute illness or abnormal vital signs (e.g.fever, SBP > 160, OR DBP > 110) per standard clinic procedures
  * The study participant understands the study and gives informed consent for participation
  * Willingness to share a positive test result for malaria or helminths with the C.H. Rennie Hospital or the Duport Road Health Center so treatment can be initiated if necessary
* For children, a study participant must satisfy the following criteria to be enrolled in this study:

  * Children 6-12 months of age at time of visit presenting for routine care at the center without acute illness or abnormal vital signs (e.g. fever) per standard clinic procedures
  * The parent or guardian understands the study and gives informed consent for participation of their child
  * Willingness of parent/guardian to share a positive test result for malaria or helminths with the C.H. Rennie Hospital or the Duport Road Health Center so treatment can be initiated if necessary

EXCLUSION CRITERIA:

* For women, prior enrollment in the study during the same pregnancy
* For children, prior enrollment in the study
* Conditions that in the judgment of the Principal Investigator or Clinical Investigators could adversely impact the safety of the study participant, including conditions that may impair the ability of the participant or participant s parent/guardian to understand the study (examples to consider may include severe acute illness at the time of enrollment, psychiatric conditio (s) that may preclude compliance with the protocol, and suspected or known drug abuse). All such exclusions and the reason for exclusion will be documented.

Min Age: 6 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Pregnant women 18 years of age and older and children 6-12 months of age presenting for routine visits at C.H. Rennie Hospital in Margibi, and Dupont Road Health Center in Monrovia.@@@
Sampling Method: Non-Probability Sample
Enrollment: 1264 (Actual)
Dates: Start 2019-10-01 (Actual); Primary Completion 2021-02-04 (Actual); Study Completion 2021-02-04 (Actual)

PRIMARY OUTCOMES:
Measurement of the frequency of P. falciparum parasitemia as defined by rapid diagnostic tests and/or blood smears | Seasonal and year of sample collection
  The frequency of P. falciparum parasitemia as defined by rapid diagnostic tests and/or blood smears

CONTACTS AND LOCATIONS:
Overall Officials: Patrick E Duffy, M.D., Principal Investigator — National Institute of Allergy and Infectious Diseases (NIAID)
Locations (2):
- Liberia (2):
  - C.H. Rennie Hospital, Margibi
  - Duport Road Health Center, Monrovia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Rogerson SJ, Desai M, Mayor A, Sicuri E, Taylor SM, van Eijk AM. Burden, pathology, and costs of malaria in pregnancy: new developments for an old problem. Lancet Infect Dis. 2018 Apr;18(4):e107-e118. doi: 10.1016/S1473-3099(18)30066-5. Epub 2018 Jan 31. PMID 29396010
- [Background] Kwan JL, Seitz AE, Fried M, Lee KL, Metenou S, Morrison R, Kabyemela E, Nutman TB, Prevots DR, Duffy PE. Seroepidemiology of helminths and the association with severe malaria among infants and young children in Tanzania. PLoS Negl Trop Dis. 2018 Mar 26;12(3):e0006345. doi: 10.1371/journal.pntd.0006345. eCollection 2018 Mar. PMID 29579050